CLINICAL TRIAL: NCT01705184
Title: Phase II Study Evaluating the Interest of the Re-introduction of Pemetrexed and Platinum (Cisplatin or Carboplatin) With Prolonged Angiogenic Blocking by Bevacizumab in Non Squamous Non Small Cell Lung Cancer of Advanced Stage.
Brief Title: Re-introduction of Pemetrexed and Cisplatin With Prolonged Angiogenic Blocking by Bevacizumab in Advanced Lung Cancer.
Acronym: BUCiL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1102; 2012-002647-18 (EudraCT Number)
Record Dates: First submitted 2012-10-05; First posted 2012-10-12 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Nonsquamous Nonsmall Cell Neoplasm of Lung
Keywords: Stop and go; Non-small cell lung cancer; Non-squamous; Bevacizumab; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Bevacizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BUCiL (Experimental): Sequence 1 : 3 cycles of cisplatin-pemetrexed-bevacizumab, then maintenance by bevacizumab if disease control. If progression --> Sequence 2
  Sequence 2 : 3 cycles of cisplatin-pemetrexed-bevacizumab, then maintenance by bevacizumab-pemetrexed if disease control
  Interventions: Drug: Cisplatin; Drug: Bevacizumab; Drug: Pemetrexed

INTERVENTIONS:
Drug: Cisplatin — 75 mg/m2, IV (in the vein) on day 1 of each 21 day cycle. During 3 cycles of each sequence
Drug: Bevacizumab — 7,5 mg/kg, IV (in the vein) on day 1 of each 21 day cycle until progression for each sequence
Drug: Pemetrexed — 500 mg/m2, IV (in the vein) on day 1 of each 21 day cycle. During 3 cycles for the 1st sequence and until progression for the 2nd sequence.

SUMMARY:
At present, the treatment of non-squamous cell lung cancer is based on chemotherapy with platinum eventually associated with bevacizumab. A new treatment begins at progression.

In colo-rectal metastatic cancer, it was demonstrated that the first-line of treatment could be administered according to a stop and go strategy respecting therapeutic breaks between sequences of identical treatment. During these therapeutic breaks, a treatment of maintenance is possibly better than an absence of treatment. These plans benefit to the patients in terms of efficiency but also in terms of toxicity, in particular neurological.

The question is to know if this strategy is feasible in lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Non squamous non small cell lung cancer histologically or cytologically confirmed with no EGFR mutation.
* Stage IV NSCLC. Patient with cerebral metastasis are eligible if the metastasis is asymptomatic.
* Measurable disease (recist criteria)
* Age ≥18 years
* PS0 or 1

Exclusion Criteria:

* Mixed cancer small cells and non small cells or squamous lung cancer . EGFR mutated cancer
* History of malignant tumour excepted cervical and basocellular cancer and cancer cured for at least 5 years.
* Tumor invaded the big vessels or the proximal visible in TDM.
* History of adjuvant or neoadjuvant chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Feasibility | After 3 cycles
  Number of patients receiving 3 cycles of chemotherapy with full-dose platinum in the 2nd sequence

SECONDARY OUTCOMES:
Control rate after the 2nd sequence | After 3 cycles
Response rate after the 1st sequence | After 3 cycles
Overall survival | 12 months
Quality of life | During Sequence 2 : at the beginning and after 3 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Jaafar BENNOUNA, MD, Principal Investigator — Centre René Gauducheau - Nantes
Locations (12):
- France (12):
  - Avignon - Institut Sainte-Catherine, Avignon
  - Caen - Centre François Baclesse, Caen
  - Caen - CHU Côte de Nacre, Caen
  - Centre Hospitalier, Chauny
  - CH du Mans, Le Mans
  - Hôpital Nord - Oncologie Multidisciplinaire & Innovations Thérapeutiques, Marseille
  - Mulhouse - CH, Mulhouse
  - Nantes - Centre René Gauducheau, Nantes
  - Hopital Tenon - Pneumologie, Paris
  - HCL - Lyon Sud (Pneumologie), Pierre-Bénite
  - Rennes - CHU, Rennes
  - Strasbourg - NHC, Strasbourg

REFERENCES:
- [Background] Tournigand C, Cervantes A, Figer A, Lledo G, Flesch M, Buyse M, Mineur L, Carola E, Etienne PL, Rivera F, Chirivella I, Perez-Staub N, Louvet C, Andre T, Tabah-Fisch I, de Gramont A. OPTIMOX1: a randomized study of FOLFOX4 or FOLFOX7 with oxaliplatin in a stop-and-Go fashion in advanced colorectal cancer--a GERCOR study. J Clin Oncol. 2006 Jan 20;24(3):394-400. doi: 10.1200/JCO.2005.03.0106. PMID 16421419
- [Background] Paz-Ares L, de Marinis F, Dediu M, Thomas M, Pujol JL, Bidoli P, Molinier O, Sahoo TP, Laack E, Reck M, Corral J, Melemed S, John W, Chouaki N, Zimmermann AH, Visseren-Grul C, Gridelli C. Maintenance therapy with pemetrexed plus best supportive care versus placebo plus best supportive care after induction therapy with pemetrexed plus cisplatin for advanced non-squamous non-small-cell lung cancer (PARAMOUNT): a double-blind, phase 3, randomised controlled trial. Lancet Oncol. 2012 Mar;13(3):247-55. doi: 10.1016/S1470-2045(12)70063-3. Epub 2012 Feb 16. PMID 22341744
- [Background] Chibaudel B, Maindrault-Goebel F, Lledo G, Mineur L, Andre T, Bennamoun M, Mabro M, Artru P, Carola E, Flesch M, Dupuis O, Colin P, Larsen AK, Afchain P, Tournigand C, Louvet C, de Gramont A. Can chemotherapy be discontinued in unresectable metastatic colorectal cancer? The GERCOR OPTIMOX2 Study. J Clin Oncol. 2009 Dec 1;27(34):5727-33. doi: 10.1200/JCO.2009.23.4344. Epub 2009 Sep 28. PMID 19786657
- See also: IFCT website — http://www.ifct.fr